CLINICAL TRIAL: NCT06448715
Title: Real-World Treatment Study of Soliris (Eculizumab)
Acronym: SolirisPMS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D7412R00001
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Observational

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
As part of a post-approval commitment, the Korean health authority requests a study to characterize safety and effectiveness in patients who are treated with Soliris in normal clinical practice settings. This study is designed to assess the known safety profile or identify previously unsuspected adverse reactions and to evaluate the effectiveness of Soliris under conditions of routine daily medical practice in Korea.

This study will provide information on the population of Korean patients who are treated with Soliris.

DETAILED DESCRIPTION:
The Korea Risk Management Plan (K-RMP) of Soliris Inj. 300mg (eculizumab, hereinafter referred to as 'Soliris' or study drug) includes Post-Marketing Surveillance (PMS) as part of the pharmacovigilance plan in accordance with 'Article 7-2 of Regulation on Pharmaceuticals Approval, Notification and Review'.

This study will be conducted to prepare data on drug use results required for post- marketing re-examination application of Soliris and the purpose of the study is to identify the safety under real world practice.

Soliris was approved by the Ministry of Food and Drug Safety on February 18, 2021 for the treatment of Neuromyelitis Optica Spectrum Disorder (NMOSD) in adult patients who are anti-aquaporin-4 (AQP-4) antibody positive, and a 4 years of re-examination period was given based on the approval date of the indication and usage change.

The re-examination period for Soliris is calculated as February 17, 2025 in accordance with the 'Standards for Re-examination of New Drugs, etc.' This study includes about 11 adult patients with NMOSD positive for anti-aquaporin-4 (AQP-4) antibody currently treated with or initiating treatment with Soliris .

It will be conducted as a total surveillance method in which each subject who received the drug is recorded in the case report form during the study period. In addition, efforts will be made to conduct investigations on safety and efficacy, such as onset of side effect and expected effects, for all patients who received the product up to two years from the marketing date.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 or older with NMOSD positive for anti-aquaporin-4 (AQP-4) antibody who are receiving or starting treatment with Soliris according to the product label
2. Patients who have been vaccinated against Neisseria meningitidis at least 2 weeks prior to receiving the first dose of Soliris. However, patients who receive Soliris within 2 weeks after Neisseria meningitidis vaccination should receive treatment with appropriate prophylactic antibiotics for 2 weeks after vaccination
3. Patient who understood and consented to the written informed consent provided.

Exclusion Criteria:

1. Patients with hypersensitivity to eculizumab, murine protein, or any other component of Soliris
2. Patients with untreated serious Neisseria meningitidis infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: According to the medical judgment of the investigator, patients who received Soliris in accordance with product label will be enrolled if they meet all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
safety assessment of soliris | 24 weeks
  Safety (adverse events (AEs), serious AEs (SAEs), adverse drug reactions (ADRs), serious ADRs (SADRs), unexpected AEs/ADRs)

SECONDARY OUTCOMES:
efficacy assessment of Soliris | 24 weeks
  relapse of NMOSD

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7412R00001&attachmentIdentifier=1b4fe60d-66cc-4120-afd7-131593ee0e67&fileName=D7412R00001_Clinical_Study_Report_(CSR)_Synopsis_Redacted.pdf&versionIdentifier=